CLINICAL TRIAL: NCT06035211
Title: Effect on Pre-operative Anxiety of a Personalized Three-dimensional Kidney Model Prior to Nephron-sparing Surgery for Renal Tumor. R3DP-A
Brief Title: Effect on Pre-operative Anxiety of a Personalized Three-dimensional Kidney Model Prior to Nephron-sparing Surgery- Rein 3D Anxiety
Acronym: R3DP-A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2022/18
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Tumoral Kidney
Keywords: Kidney Neoplasms; Renal-Cell Carcinoma; Nephron-Sparing Surgery; 3D Modeling; 3D Printing; Anxiety; STAI; Personalized Medicine
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual 3D model group (Active Comparator): exchange time with the virtual 3D model of the kidney to be operated on as information support
  Interventions: Other: 3D model pré-operative education
- 3D Printed Model Group (Active Comparator): eexchange time with the printed three-dimensional model of the kidney to be operated on as information support
  Interventions: Other: 3D model pré-operative education
- Control group (No Intervention): discussion time with the patient information sheet of the French Association of Urology (AFU) as information support

INTERVENTIONS:
Other: 3D model pré-operative education — Before surgery, during a preoperative therapeutic education consultation, 3D models will be presented to the patients according to the allocated study group
  Arms: 3D Printed Model Group; Virtual 3D model group

SUMMARY:
The goal of this clinical trial is to evaluate the impact of showing and handling a three-dimensional modelization of a patient's tumoral kidney the day before his nephron-sparing surgery. The main outcome measure was the effect on anxiety assessed via the STAI state score. 3 types of pre-operative information were compared (3D virtual model, 3D printed model, and information) using a randomization.

DETAILED DESCRIPTION:
Announcement of serious illnesses and especially cancerous disease has major impacts on one's psychological field. Need of surgery can create even other fears due to its unknown nature. Use of tools to decrease anxiety and enhance understanding prior to surgery is a key point in comprehensive care that is way not enough promoted for now. In the field of surgery, available methods to deal with pre-operative anxiety are massively represented by anxiolytics drugs, only few other devices were evaluated.

Technological development in healthcare has seen the rising of three-dimensional media, especially in surgery, for procedure planning. There is no doubt that this tool is effective in helping surgeons regarding the studies published within the past few years but there is no such evidence concerning the benefit for patients. Some authors report improvement of patients understanding and great satisfaction referring to the usefulness of this tool. But none of these papers evaluated anxiety.

The goal of this research is to measure the effect of a personalized three-dimensional model of patients' tumoral kidney on peri-operative anxiety.

For this purpose this clinical trial is designed as following: a total of 234 (78*3) patients planned to have a nephron-sparing surgery for kidney tumor are going to be randomly assign in 3 different groups. Inside the 2 interventional groups, patients' kidneys will be modelled in three dimensions, but in one of the two groups, the model will be 3D-printed. The control group will include patients for whom the pre-operative information will be made based on standardized information letter from the French Urological Association.

Before surgery, during a preoperative therapeutic education consultation, 3D models will be presented to the patients according to the allocated study group. All patients will have to complete questionnaires to assess their anxiety level, their quality of life, their health literacy level and their understanding of disease and surgical procedure.

One month after surgery, during the post-operative consultation, patients will also fill out the different questionnaires to assess their anxiety level, quality of life, and level of litteracy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age)
* Scheduled surgical management by laparoscopic partial nephrectomy with robotic assistance for kidney tumor
* Unilateral kidney tumor or 1st surgery for bilateral involvement
* Consent expressed for integration of the UroCCR cohort,
* Expressed consent for participation in the 3D Anxiety study.
* Patients affiliated or benefiting from a social security plan

Exclusion Criteria:

* Refusal of consent or participation
* Difficulty understanding and expressing oneself in French
* Patient under guardianship or curatorship
* No preoperative CT scan available for 3D modeling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-09-19 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the mean pre-operative anxiety score per arm, by filling the STAI-state self-questionnaire | Day-1 from surgery
  The STAI-Etat will be collected before surgery to evaluate the effect of using a personalized three-dimensional model of the patient's kidney during a pre-operative information visit .

SECONDARY OUTCOMES:
Measurement of the progression of the mean anxiety score per arm, by filling STAI-Trait Anxiety self-questionnaire. | between baseline and Day 15 post-op
  The progression of the mean anxiety score per arm, measured by STAI-State self-questionnaire at the three follow-up visits in the study and adjusted on the STAI-Trait score at baseline will assess feelings of apprehension, tension, nervousness and worries that the subject usually feels.
Measurement of the progression in mean health literacy questionnaire score HLSEU-Q16 between baseline and 15-day post-operative follow-up per arm | between baseline and Day 15 post-op
  This questionnaire is a short version version of the European Health Literacy Survey Questionnaire based on a model including 4 health information processing skills: accessing, understanding, evaluating and applying application of health information .
Measurement of the mean pre-operative score for understanding disease and choice of treatment per arm by filling the WAKE questionnaire | Day-1 from surgery
  The WAKE questionnaire is used assess the feeling of understanding of the disease and the choice of treatment preoperatively in each of the three groups, the questionnaire comprises five question on the understanding of the disease . Each dimension has 5 levels : very poor, poor,faire, good, very good or strongly desagree, disagree,neutral,agree or strongly agree
Measurement of the progression of quality of life in each of the three groups by filling the EQ-5D-5L questionnaire | between inclusion and Day 15 post-op
  The EQ-5D-5L questionnaire measures participants' quality of life.The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Additinonally, the questionnaire records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Measurement of the average duration of the pre-operative information visit in each of the three groups | between Day-21 and Day-4 from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe BERNHARD, Professeur, Principal Investigator — University Hospital, Bordeaux
Locations (6):
- France (6):
  - CHU d'ANGERS, Angers
  - CHU de Bordeaux, Bordeaux
  - CHU de CAEN, Caen
  - Hôpital Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - CHU de La CONCEPTION, Marseille
  - CHU de NANTES, Nantes